CLINICAL TRIAL: NCT07371234
Title: A Single Arm, Phase II Clinical Study of Low-Dose Radiotherapy Combined With Anti-PD-1 Monoclonal Antibody Immunotherapy as Neoadjuvant Treatment for Surgically Resectable, Locally Advanced Head and Neck Squamous Cell Carcinoma (HNSCC)
Brief Title: Low-Dose Radiotherapy and Anti-PD-1 Immunotherapy as Neoadjuvant Treatment for Resectable Locally Advanced Head and Neck Squamous Cell Carcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Xiwei XU (Other)
Responsible Party: Sponsor-Investigator, Xiwei XU, Attending Physician, Fifth Affiliated Hospital, Sun Yat-Sen University
Organization: Fifth Affiliated Hospital, Sun Yat-Sen University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZDWY.FSZLK.011
Record Dates: First submitted 2026-01-19; First posted 2026-01-27 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Locally Advanced Head and Neck Squamous Cell Carcinoma
Keywords: low-dose radiotherapy; neoadjuvant immunotherapy; Locally Advanced Head and Neck Squamous Cell Carcinoma
MeSH Terms: interventions — Neoadjuvant Therapy; Radiotherapy; Surgical Procedures, Operative; Radiotherapy, Adjuvant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Low-Dose RT plus Anti-PD-1 Imunotherapy Arm (Experimental): Patients receive low-dose radiotherapy combined with anti-PD-1 monoclonal antibody immunotherapy as neoadjuvant treatment prior to surgical resection.
  Interventions: Drug: Neoadjuvant and Adjuvant Immunotherapy; Radiation: Low-dose radiotherapy; Procedure: Surgery; Radiation: Adjuvant Radiotherapy; Drug: Adjuvant Cisplatin

INTERVENTIONS:
Drug: Neoadjuvant and Adjuvant Immunotherapy — Neoadjuvant therapy with Toripalimab (240mg, Day 1, Q3W, 2 cycles);Adjuvant immunotherapy with Toripalimab (240mg, Day 1, Q3W, for a total of 15 cycles).
Radiation: Low-dose radiotherapy — Low-dose radiotherapy (1 Gy/fraction, on Days 1, 8, and 15 of each cycle, Q3W, for 2 cycles; total dose: 6 Gy in 6 fractions).
Procedure: Surgery — Radical surgery performed 3-4 weeks after neoadjuvant therapy, following a re-evaluation of surgical indications by the surgeon.
Radiation: Adjuvant Radiotherapy — Low-risk group: 60 Gy in 30 fractions, using intensity-modulated radiation therapy (IMRT); High-risk group: 66 Gy in 33 fractions, or 70 Gy in 35 fractions for residual lesions, using intensity-modulated radiation therapy (IMRT).
Drug: Adjuvant Cisplatin — High-risk group：Cisplatin 100 mg/m² is administered via intravenous infusion on Day 1 of every 21-day cycle during radiotherapy, for a total of 3 cycles.

SUMMARY:
Over 60% of head and neck squamous cell carcinoma (HNSCC) patients are diagnosed at a locally advanced stage. While standard treatments involve surgery and chemoradiotherapy, prognosis remains poor, with 50-60% experiencing local recurrence within two years. Neoadjuvant therapy can potentially reduce tumor burden, preserve organs, and lower distant metastasis risk. Despite the KEYNOTE-689 trial showing that adjuvant two-cycle pembrolizumab increased major pathological response to 9.8% in stage III-IVB HNSCC, this result remains insufficient. More effective immunotherapy-based combinations are urgently needed to improve long-term survival after neoadjuvant treatment.

Preclinical and clinical evidence indicates that low-dose radiotherapy can activate the tumor immune microenvironment and synergize with immunotherapy. Based on this rationale, the present clinical trial will evaluate a neoadjuvant regimen combining LDRT with two cycles of an anti-PD-1 inhibitor in patients with surgically resectable, locally advanced HNSCC.

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily sign and date the informed consent form.
* Untreated, histologically confirmed squamous cell carcinoma of the head and neck (oral cavity, oropharynx, hypopharynx, or larynx) with CPS ≥1, classified as stage T3-4bN0M0 or T1-4bN1-3M0, corresponding to stage III-IVB according to the AJCC Staging System, 8th Edition.
* Deemed eligible for curative surgery based on surgeon's assessment.
* Age: 18 to 75 years.
* ECOG performance status of 0 or 1.
* Life expectancy greater than 6 months.
* At least one measurable lesion as per RECIST 1.1 criteria.
* Adequate organ function, defined as meeting all the following criteria (without receipt of blood products, colony-stimulating factors, or hematopoietic growth factors within 14 days prior to testing): Hemoglobin ≥ 90 g/L Absolute neutrophil count ≥ 1.5 × 10⁹/L Platelet count ≥ 100 × 10⁹/L Serum albumin ≥ 28 g/L Total bilirubin ≤ 1.5 × upper limit of normal (ULN) ALT and AST ≤ 2.5 × ULN Serum creatinine ≤ 1.5 × ULN or creatinine clearance ≥ 50 mL/min Activated partial thromboplastin time (aPTT) and international normalized ratio (INR) ≤ 1.5 × ULN (patients on a stable dose of anticoagulant therapy such as low molecular weight heparin or warfarin are eligible if INR is within the therapeutic range) Thyroid-stimulating hormone (TSH) ≤ ULN; if abnormal, T3 and T4 levels must be evaluated, and patients with normal T3 and T4 levels are eligible.
* Women of childbearing potential must agree to use effective contraception (e.g., intrauterine device, oral contraceptives, or condoms) during the treatment period and for 3 months after the last dose.
* Good compliance with the study protocol.

Exclusion Criteria:

* Pregnant or lactating women.
* History of allergy to PD-1 inhibitors.
* History of other malignancies within the past 5 years or at the time of enrollment, with the exception of cured basal cell carcinoma of the skin, carcinoma in situ of the cervix, and papillary thyroid carcinoma.
* Uncontrolled cardiac clinical symptoms or diseases, such as: (1) heart failure of NYHA Class II or higher, (2) unstable angina, (3) myocardial infarction within the past year, and (4) patients with clinically significant ventricular or supraventricular arrhythmias requiring intervention.
* Any of the following prior treatments: ① Receipt of any investigational drug prior to the first dose of the current study drug. ② Concurrent participation in another clinical study, unless it is an observational (non-interventional) study or an interventional study during the follow-up phase. ③ Systemic treatment with corticosteroids (>10 mg prednisone daily or equivalent) or other immunosuppressive agents within 2 weeks prior to the first dose of the study drug, with the exception of topical corticosteroid use for local inflammation, prevention of allergic reactions, or management of nausea and vomiting. Inhaled or topical steroids and physiologic replacement doses of corticosteroids (≤10 mg prednisone equivalent daily) are permitted in the absence of active autoimmune disease. ④ Administration of live vaccines within 4 weeks prior to the first dose of the study drug. ⑤ Major surgery or severe trauma within 4 weeks prior to the first dose of the study drug.
* Severe infection (Grade >2 according to Common Terminology Criteria for Adverse Events), such as severe pneumonia, bacteremia, or complicating infections requiring hospitalization, occurring within 4 weeks prior to the first dose of the study drug; or active pulmonary inflammation or signs/symptoms of infection indicated by baseline chest imaging within 2 weeks prior to the first dose, or requiring oral or intravenous antibiotic treatment (excluding prophylactic antibiotics).
* History of active autoimmune diseases and syndromes (including but not limited to interstitial pneumonia, colitis, hepatitis, hypophysitis, vasculitis, nephritis, hyperthyroidism, and hypothyroidism). Patients with vitiligo not requiring intervention in adulthood, or childhood asthma/allergies that have resolved, are not excluded.
* History of immunodeficiency, including HIV positivity, other acquired or congenital immunodeficiency diseases, or history of organ or bone marrow transplantation.
* Patients with active tuberculosis infection based on medical history or CT findings, or a history of active tuberculosis infection within 1 year prior to enrollment, or a history of active tuberculosis infection more than 1 year ago without adequate course of anti-tuberculosis therapy.
* Active hepatitis B (HBV DNA ≥ 2,000 IU/mL or 10,000 copies/mL) or hepatitis C (positive HCV antibody test with HCV RNA above the lower limit of detection).
* Known history of substance abuse, alcohol abuse, or drug use.
* Considered ineligible for participation based on the investigator's judgment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2025-12-15 (Actual); Primary Completion 2027-01-15 (Estimated); Study Completion 2028-12-30 (Estimated)

PRIMARY OUTCOMES:
Main pathological response rate | 1 week post-surgery
  The proportion of patients with residual living tumor cells in the tumor bed under microscopy after HE staining of the specimens organized is less than 10%.

SECONDARY OUTCOMES:
Progression-free survival | 2 years after enrollment treatment
  From random grouping to the time interval until tumor progression or death for any reason, or until the last follow-up time if there is no tumor progression.
Pathological complete response rate | 1 week post-surgery
  The proportion of patients with no residual live tumor cells under the microscope.
Objective response rate | 3-4 weeks after neoadjuvant therapy
  Evaluate the proportion of patients with objective response (complete response and partial response) through imaging assessments such as MRI and CT.
Overall survival | 2 years after enrollment treatment
  The time interval from random grouping to the time of death for any reason, or to the last follow-up time if there is no death.
Adverse Events Reporting | 1 year
  Number of participants with treatment-related adverse events as assessed by CTCAE v5.0
Head and Neck Cancer-Specific Quality of Life | 1 year
  Changes from baseline in head and neck cancer-specific symptoms and functions were assessed using the EORTC QLQ-H&N35 module (European Organization for Research and Treatment of Cancer Quality of Life Questionnaire, Head and Neck Cancer Module). The scores range from 0 to 100, with higher scores indicating a better quality of life outcome and lower scores indicating worse symptoms or functions.
Health-related Quality of Life | 1 year
  Changes from baseline in patient-reported quality of life were assessed using the EORTC QLQ-C30 (European Organization for Research and Treatment of Cancer Quality of Life Questionnaire, Version 3.0). The scores range from 0 to 100, with higher scores indicating a better quality of life outcome and lower scores indicating worse symptoms or functions.
Pathological tumor remission rate -2 | 1 week post-surgery
  The proportion of patients with tumor necrosis under a microscope, where the ratio of keratin fragments and giant cells/tissue cells in tissue sections is not less than 50%.
Non-surgical delay rate | 8 weeks after two cycles of neoadjuvant therapy
  The proportion of patients whose surgical time is more than 4 weeks longer than planned.
R0 resection rate | 1 week post-surgery
  The proportion of patients who achieved R0 resection (where the tumor is completely excised during surgery and the margin tissue pathology is negative) among all patients who underwent surgical resection.

CONTACTS AND LOCATIONS:
Overall Officials: Rui You, Study Director — The Fifth Affiliated Hospital, Sun Yat-sen University
Locations (1):
- The Fifth Affiliated Hospital,Sun Yat-sen University, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided